CLINICAL TRIAL: NCT01495065
Title: A Two Part Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of GSK2251052 After Single Ascending Dosesand Repeat Doses of IV GSK2251052 in Healthy Male Japanese and Caucasian Subjects and a Repeat Dose Study to Evaluatesupratherapeutic Doses of IV GSK2251052 in Healthy Volunteers
Brief Title: A Study to Evaluate Single and Repeat Doses of IV GSK2251052 in Healthy Male Japanese and Caucasian Subjects and Repeat Doses of Supratherapeutic Doses of IV GSK2251052 in Healthy Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 116160
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Community-acquired Infection
Keywords: GSK2251052, healthy volunteer, safety, tolerability, pharmacokinetics, single
MeSH Terms: conditions — Community-Acquired Infections | interventions — 3-(aminomethyl)-7-(3-hydroxypropoxy)-1-hydroxy-1,3-dihydro-2,1-benzoxaborole; BID protein, human; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Part A (Experimental): Japanese subjects in cohort 1 and 2 will receive treatments A, B and C. Caucasian subjects in cohort 3 will receive treatment B and C.
  Interventions: Drug: GSK2251052 750 mg; Drug: GSK2251052 1500 mg; Drug: GSK2251052 1500 mg BID
- Part B (Experimental): Subjects in cohort 4 and 5 will receive repeat doses of IV GSK2251052 for 10 days.
  Interventions: Drug: GSK2251052 2250 mg; Drug: GSK2251052 3000 mg; Drug: GSK2251052 0.9% saline

INTERVENTIONS:
Drug: GSK2251052 750 mg — Treatment A: 750 mg IV GSK2251052 single dose
  Arms: Part A
Drug: GSK2251052 1500 mg — Treatment B: 1500 mg IV GSK2251052 single dose
  Arms: Part A
Drug: GSK2251052 1500 mg BID — Treatment C: 1500 mg IV GSK2251052 BID or placebo for 12 days
  Arms: Part A
Drug: GSK2251052 2250 mg — Treatment D: On Day 1 a single dose of GSK2251052 2250 mg IV administered over 60 minutes; Days 4 - 12 BID doses of GSK2251052 2250 mg IV (for 9 days), fasted
  Arms: Part B
Drug: GSK2251052 3000 mg — Treatment E: On Day 1 a single dose of GSK2251052 3000 mg IV administered over 60 minutes; Days 4 - 12 BID doses of GSK2251052 3000mg IV (for 9 days), fasted
  Arms: Part B
Drug: GSK2251052 0.9% saline — Treatment P: On Day 1 a single dose of 0.9% saline IV administered over 60 minutes; On Days 4 - 12 BID doses of 0.9% saline (for 9 days), fasted
  Arms: Part B

SUMMARY:
This is a two-part study. Part A is a three-period study in approximately 24 healthy male Japanese and Caucasian subjects. Period 1 and Period 2 will be an open label study to investigate the safety, tolerability, and pharmacokinetics of single ascending intravenous doses of GSK2251052. Period 3 is a single blind, placebo controlled, repeat fixed dose design to evaluate the safety, tolerability and pharmacokinetics of multiple intravenous doses of GSK2251052 for 12 days. The selection of the repeat IV dose will be based on the results from Periods 1 and 2. Japanese subjects will be stratified based on their metabolic genotype, polymorphic or wild-type for ADH and ALDH. Caucasian subjects are not anticipated to have these enzyme polymorphisms and therefore will not be stratified.

Part B is a two cohort, single-blind, randomized, placebo-controlled, dose-rising, repeat dose study in approximately 24 healthy male and female subjects to evaluate the safety, tolerability, and pharmacokinetics of supratherapeutic IV doses of GSK2251052 for 10 days. Cohort 1 subjects will be randomized to receive 2250 mg of GSK2251052 or placebo and Cohort 2 subjects will be randomized to receive 3000 mg GSK2251052 or placebo. The decision to conduct Cohort 2 of Part B will be based on the available toxicology cover results from ongoing preclinical toxicity studies.

ELIGIBILITY:
Inclusion Criteria:

* AST, ALT, alkaline phosphatase and bilirubin ≤ 1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Healthy adult male Japanese or healthy adult Caucasian male. In Part B, healthy adult males or females (Part B only) as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters outside the reference range for the population being studied may be included only if the Investigator and the GSK Medical Monitor agree that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures. Subjects with coagulation, reticulocyte, or Hgb values outside the normal range should always be excluded from enrollment.
* Japanese defined as being born in Japan, having four ethnic Japanese grandparents, holding a Japanese passport or identity papers and being able to speak Japanese. Japanese subjects should also have lived outside Japan for less than 10 years.
* The following genetic variants of ADH and ALDH will be acceptable: Group 1 Japanese: ADH1B (*/1*1), ADH1B (*1/*2), ADH1B (*2/*2); ALDH2 (*1/*1). Group 2 Japanese: ADH1B (*/1*1), ADH1B (*1/*2), ADH1B (*2/*2); ALDH2 (*1/*2); ADH1B (*/1*1), ADH1B (*1/*2), ADH1B (*2/*2); ALDH2 (*2/*2). Group 3 Caucasian: ADH1B (*/1*1); ALDH2 (*1/*1)
* Part A: Japanese or Caucasian Male between 20 and 65 years of age inclusive, at the time of signing the informed consent. Part B: Males or Females between 18 and 55 years of age inclusive, at the time of signing the consent.
* Male subjects with female partners of child-bearing potential must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until 21 days after the final dose.
* A female is eligible to enter and participate in this study if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant), including any female who: Has had a hysterectomy or Has had a bilateral oophorectomy (removal of the ovaries) or Has had a bilateral tubal ligation or Is post-menopausal (a demonstration of total cessation of menses for ≥ 1 year from the date of screening visit). A follicle stimulating hormone (FSH) level will be performed to confirm a post-menopausal state. For this study FSH levels ≥ 40mIU/mL are consistent with menopause. If a subject is on estrogen replacement and menopausal status is questionable, estrogen replacement should be discontinued for 2 weeks and then the subject rescreened, as estrogen replacement can suppress FSH.
* Part A: For Japanese subjects: Body weight ≥ 50 kg and BMI within the range 18.5 - 29.0 kg/m2 (inclusive). For Caucasian subjects: Body weight ≥ 50 kg and BMI within the range 19 - 32 kg/m2 (inclusive). Part B: Body weight ≥ 50 kg for males and 45 kg for females and BMI within the range 18.5- 31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.
* QTc, QTcB or QTcF < 450 msec; or QTc < 480 msec in subjects with Bundle Branch Block.

Exclusion Criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study.
* History of bleeding or clotting disorders including disseminated intravascular coagulation, hemophilia Henoch-Schönlein purpura (allergic purpura), hereditary hemorrhagic telangiectasia, thrombocytopenia, thrombophilia or Von Willebrand's disease.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* A positive pre-study drug/alcohol screen.
* History of regular alcohol consumption within 6 months of the study defined as: an average weekly intake of >14 drinks for males or >7 drinks for females. One drink is equivalent to 12 g of alcohol: 12 ounces (360 ml) of beer, 5 ounces (150 ml) of wine or 1.5 ounces (45 ml) of 80 proof distilled spirits.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Part A: Female subjects. Part B: Female subjects of child-bearing potential. Unwillingness or inability to follow the procedures outlined in the protocol.
* Subject is mentally or legally incapacitated.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Unwilling to abstain from alcohol for at least 7 days prior to dose until 21 days after the final dose of study medication.
* Part A: Subjects with a smoking history of >10 cigarettes per day in the last 3 months. Part B: History or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* Subjects with a creatinine clearance < 80 mL/min as calculated by the Cockcroft- Gault equation.[Cockcroft, 1976] CLcr (mL/min) = (140 - age) * Wt / (72 * Scr) (times 0.85 if female) where age is in years, weight (Wt) is in kg, and serum creatinine (Scr) is in units of mg/dL.
* Consumption of red wine, seville oranges, grapefruit or grapefruit juice and pomelos, exotic citrus fruits, grapefruit hybrids or fruit juices from 7 days prior to the first dose of study medication.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects.
* A recent history of symptomatic orthostatic hypotension
* History of clinically significant cardiovascular disease including: Exclusion criteria for screening ECG (a single repeat is allowed for eligibility determination): Heart rate (males) <45 and >100 bpm; heart rate (females) <50 and >100 bpm. PR interval <120 and >220 msec. QRS duration <70 and >120 msec. QTc interval (Bazett) >450 msec (> 480 msec for BBB); Evidence of previous myocardial infarction (pathologic Q waves, S-T segment changes (except early repolarization); History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease; Any conduction abnormality (including but not specific to left or right complete bundle branch block, AV block [2nd degree (type II) or higher], Wolf Parkinson White [WPW] syndrome); Sinus pauses > 3 seconds; Any significant arrhythmia which, in the opinion of the principal Investigator and GSK Medical Monitor, will interfere with the safety for the individual subject.Non-sustained (≥3 consecutive ventricular ectopic beats) or sustained ventricular tachycardia.
* Subject who may be compromised by a major drop in hemoglobin and is unwilling to receive a blood transfusion if clinically indicated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-12-19 (Actual); Primary Completion 2012-02-17 (Actual); Study Completion 2012-02-17 (Actual)

PRIMARY OUTCOMES:
Composite (or Profile) of Pharmacokinetics | Part A: Period 1 for 168 hours post dose; Period 2 for 336 hours post dose; Period 3 on day 12 for 12 hours post dose. Part B: On day 1 for 72 hours post dose; on day 12 for 12 hours post dose.
  pharmacokinetic endpoints maximum observed concentration fixed nominal time (Cmax), area under the concentration-time curve from time zero extrapolated to infinite time (AUC(0-∞), area under the concentration-time curve from time zero to last time of quantifiable concentration within a subject across all treatments (AUC(0-t), AUC(0-12), time of occurrence of Cmax (tmax), time of last quantifiable concentration (tlast), terminal phase half-life (t1/2), volume of distribution at steady state (Vss), and Systemic clearance of parent drug (CL) of GSK2251052 and metabolite M3 (as appropriate).
Safety and tolerability parameters including change from baseline measures for vital signs | Part A: for 15 weeks. Part B: for 9 weeks
Safety and tolerability parameters including change from baseline for ECGs | Part A: for 15 weeks. Part B: for 9 weeks
Safety and tolerability parameters including change from baseline for clinical laboratory tests | Part A: for 15 weeks. Part B: for 9 weeks
  hematology, chemistry, and urinalysis
Safety and tolerability parameters including change from baseline in the collection of adverse events | Part A: for 15 weeks. Part B: for 9 weeks

SECONDARY OUTCOMES:
Composite (or Profile) of Pharmacokinetics | Part A: Period 1 for 168 hours post dose; Period 2 for 336 hours post dose; Period 3 on day 12 for 12 hours post dose. Part B: On day 1 for 72 hours post dose; on day 12 for 12 hours post dose.
  Observed accumulation based on (AUC(Ro) and Cmax (RCmax) and determine the steady-state ratio (Rss)
Composite or Profile of Pharmacokinetics | Part A: Period 1 for 168 hours post dose; Period 2 for 336 hours post dose; Period 3 on day 12 for 12 hours post dose. Part B: On day 1 for 72 hours post dose; on day 12 for 12 hours post dose.
  AUC(0-∞), AUC(0-t), and Cmax following IV administration at different doses for the assessment of dose proportionality

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Glendale, California, United States

REFERENCES:
- See also: Results for study 116160 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116160?search=study&search_terms=116160#rs